CLINICAL TRIAL: NCT02605005
Title: The Impact of a Beach Chair Position During Shoulder Arthroscopy on Regional Cerebral Oxygen Saturation : Comparison of Interscalene Block and General Anesthesia
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 25-1:5484-3/2013.
Record Dates: First submitted 2015-11-06; First posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Impaired Oxygen Delivery; Cerebral Hypoxia
Keywords: interscalene block, general anesthesia, shoulder arthroscopy, cerebral oxygen saturation, beach chair position
MeSH Terms: conditions — Hypoxia, Brain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GA: general anesthesia
- ISB: interscalene block

SUMMARY:
The aim of this study is to investigate the relationship between the patient positioning in the beach chair position with consequential arterial pressure changes and their influence on regional cerebral oxygen saturation under two anesthesia techniques, general anesthesia in one group of patients and interscalene block in the second group of patients.

DETAILED DESCRIPTION:
The participants of the study are patients scheduled for elective shoulder athroscopy. The patients randomise themselves by choosing the type of anesthesia technique (general anesthesia or interscalene block) after detailed description of both techniques. They receive the standard, routine medical care (monitoring and anesthesia techniques) during which the obtained data of arterial pressure, heart rate, peripheral and cerebral oxygen saturation will be statistically analysed and compared.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criterion for the study was the approval for surgery under general or regional anesthesia with ASA I and ASA II patients classification. -

Exclusion Criteria:

* The patients who have refused to take part in the study, patients assessed as ASA III or higher, who have cerebrovascular or coronary disease, coagulopathy, hypersensitivity to local anesthetics or other contraindications to one or the other type of anesthetic techniques All patients in whom the operation lasted less than 20 minutes or longer than 90 minutes, have been also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients for elective arthroscopy of the shoulder
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
changes in arterial pressure from baseline | baseline, during the operation, one hour after the operation

SECONDARY OUTCOMES:
changes in regional cerebral oxygen saturation from baseline | baseline, during the operation, one hour after the operation